CLINICAL TRIAL: NCT03604445
Title: An Open-label, Phase I Trial to Determine the Maximum-tolerated Dose and Investigate Safety, Pharmacokinetics and Efficacy of BI 905677 Administered Intravenously in Patients With Advanced Solid Tumours
Brief Title: This Study Aims to Find and Test a Safe Dose of BI 905677 in Patients With Different Types of Cancer (Solid Tumours)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1401-0001; 2017-002945-31 (EudraCT Number)
Record Dates: First submitted 2018-07-20; First posted 2018-07-27 (Actual); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2023-07

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- BI 905677 0.05 mg/kg (Experimental): 0.05 milligrams (mg) per kilogram (kg) solution for infusion BI 905677 were administered intravenously on Day 1 of each 3-week treatment cycle. Patients may continue on treatment for unlimited cycles, until disease progression or other criteria for stopping treatment are met.
  Interventions: Drug: BI 905677
- BI 905677 0.1 mg/kg (Experimental): 0.1 milligrams (mg) per kilogram (kg) solution for infusion BI 905677 were administered intravenously on Day 1 of each 3-week treatment cycle. Patients may continue on treatment for unlimited cycles, until disease progression or other criteria for stopping treatment are met.
  Interventions: Drug: BI 905677
- BI 905677 0.2 mg/kg (Experimental): 0.2 milligrams (mg) per kilogram (kg) solution for infusion BI 905677 were administered intravenously on Day 1 of each 3-week treatment cycle. Patients may continue on treatment for unlimited cycles, until disease progression or other criteria for stopping treatment are met.
  Interventions: Drug: BI 905677
- BI 905677 0.4 mg/kg (Experimental): 0.4 milligrams (mg) per kilogram (kg) solution for infusion BI 905677 were administered intravenously on Day 1 of each 3-week treatment cycle. Patients may continue on treatment for unlimited cycles, until disease progression or other criteria for stopping treatment are met.
  Interventions: Drug: BI 905677
- BI 905677 0.8 mg/kg (Experimental): 0.8 milligrams (mg) per kilogram (kg) solution for infusion BI 905677 were administered intravenously on Day 1 of each 3-week treatment cycle. Patients may continue on treatment for unlimited cycles, until disease progression or other criteria for stopping treatment are met.
  Interventions: Drug: BI 905677
- BI 905677 1.6 mg/kg (Experimental): 1.6 milligrams (mg) per kilogram (kg) solution for infusion BI 905677 were administered intravenously on Day 1 of each 3-week treatment cycle. Patients may continue on treatment for unlimited cycles, until disease progression or other criteria for stopping treatment are met.
  Interventions: Drug: BI 905677
- BI 905677 2.4 mg/kg (Experimental): 2.4 milligrams (mg) per kilogram (kg) solution for infusion BI 905677 were administered intravenously on Day 1 of each 3-week treatment cycle. Patients may continue on treatment for unlimited cycles, until disease progression or other criteria for stopping treatment are met.
  Interventions: Drug: BI 905677
- BI 905677 2.8 mg/kg (Experimental): 2.8 milligrams (mg) per kilogram (kg) solution for infusion BI 905677 were administered intravenously on Day 1 of each 3-week treatment cycle. Patients may continue on treatment for unlimited cycles, until disease progression or other criteria for stopping treatment are met.
  Interventions: Drug: BI 905677
- BI 905677 3.6 mg/kg (Experimental): 3.6 milligrams (mg) per kilogram (kg) solution for infusion BI 905677 were administered intravenously on Day 1 of each 3-week treatment cycle. Patients may continue on treatment for unlimited cycles, until disease progression or other criteria for stopping treatment are met.
  Interventions: Drug: BI 905677

INTERVENTIONS:
Drug: BI 905677 — Solution for infusion

SUMMARY:
This study is open to adults with different types of advanced cancer (solid tumours). This study is open to people in whom previous treatments were not successful. The purpose of this study is to find out the highest dose of BI 905677 the participants can tolerate. BI 905677 is a type of an antibody that is being developed to treat cancer.

One dose of BI 905677 is given to the participants every 2 or 3 weeks as infusion into a vein. In this study, BI 905677 is given to humans for the first time. The participants visit the study site at least once a week so that the doctors can check their general health. The participants are in the study for as long as they benefit from and can tolerate treatment.

ELIGIBILITY:
Inclusion criteria

* Histologically or cytologically confirmed diagnosis of an advanced, unresectable and/or metastatic non-haematologic malignancy. Patient must have measurable or evaluable lesions (according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1).
* Patient who has failed conventional treatment or for whom no therapy of proven efficacy exists or who is not eligible for established treatment options. Patient must have exhausted treatment options known to prolong survival for their disease.
* Patient willing to undergo mandatory skin biopsy at the timepoints specified in the protocol.
* Eastern Cooperative Oncology Group score of 0 or 1.
* Adequate organ function defined as all of the following:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L; haemoglobin ≥ 9.0 g/dL; platelets ≥ 100 x 109/L without the use of hematopoietic growth factors within 4 weeks of start of study medication.
  * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN), except for patients with Gilbert's syndrome: total bilirubin ≤ 3 x ULN or direct bilirubin ≤ 1.5 x ULN.
  * Creatinine ≤ 1.5 x ULN. If creatinine is > 1.5 x ULN, patient is eligible if concurrent creatinine clearance ≥ 50 ml/min (measured or calculated by CKDEPI formula or Japanese version of CKD-EPI formula for Japanese patients).
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 x ULN if no demonstrable liver metastases, or otherwise ≤ 5 x ULN
  * Alkaline Phosphatase < 5 x ULN
* Recovered from any previous therapy-related toxicity to ≤ Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at start of treatment (except for alopecia and stable sensory neuropathy which must be ≤ CTCAE Grade 2).
* At least 18 years of age at the time of consent or over the legal age of consent in countries where that is greater than 18 years.
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
* Life expectancy ≥ 3 months at the start of treatment in the opinion of the investigator.
* Male or female patients. Women of childbearing potential (WOCBP) must only be included after a confirmed menstrual period within the past 4 weeks and a negative pregnancy test at screening. WOCBP with irregular menstruation may be included after two negative pregnancy tests during screening between 2 and 4 weeks apart. WOCBP and men who are able to father a child must be ready and able to use highly effective methods of birth control, per ICH M3 (R2), that result in a low failure rate of less than 1% per year when used consistently and correctly. These methods must be used during the study and for at least 6 months after the last dose of BI 905677. A list of contraception methods meeting these criteria is provided in the patient information.

Exclusion criteria

* Major surgery (major according to the investigator's assessment) performed within 4 weeks prior to first trial treatment or planned within 6 months after screening.
* Previous or concomitant malignancies other than the one treated in this trial within the last 2 years, except;

  * effectively treated non-melanoma skin cancers
  * effectively treated carcinoma in situ of the cervix
  * effectively treated ductal carcinoma in situ
  * other effectively treated malignancy that is considered cured by local treatment
* Osteoporosis ≥ Common Terminology Criteria for Adverse Events (CTCAE) Grade 2
* Chronic corticosteroid use
* Osteoporotic compression fracture within 12 months prior to informed consent which is clinically significant in the opinion of the investigator.
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
* Previous treatment in this trial.
* Treatment with a systemic anti-cancer therapy or investigational drug within 28 days or 5 half-lives (whichever is shorter) of the first treatment with the study medication.
* Any history of or concomitant condition that, in the opinion of the investigator, would compromise the patient's ability to comply with the study or interfere with the evaluation of the safety and efficacy of the test drug.
* Women who are pregnant, nursing, or who plan to become pregnant or nurse during the trial or within 6 months after the last dose of study treatment.
* Active alcohol or drug abuse in the opinion of the investigator.
* Patient unwilling or unable to comply with the protocol.
* Presence or history of uncontrolled or symptomatic brain or subdural metastases, unless considered stable by the investigator and local therapy was completed. Inclusion of patients with newly identified brain metastasis/es at screening will be allowed if patients are asymptomatic.
* Known history of human immunodeficiency virus (HIV) infection or an active hepatitis B or C infection which in the opinion of the investigator may interfere with participation in the trial.
* History of severe hypersensitivity reactions to monoclonal antibodies.
* History of allergy to kanamycin or similar class drugs (including streptomycin, gentamicin, amikacin, tobramycin and neomycin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - University of Southern California, Los Angeles, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York
- National Cancer Center Hospital East, Chiba, Kashiwa, Japan
- Erasmus MC Kanker Instituut, Rotterdam, Netherlands
- Hospital Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-randomised, open-label, single arm, dose escalation trial was planned to determine the maximum tolerated dose (MTD) of BI 905677 given as an intravenous infusion and to determine the recommended dose and dosing schedule for further trials in the development of BI 905677. Two treatment schedules (A and B) were planned. But only Schedule A was conducted.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 905677 0.05 mg/kg: 0.05 milligrams (mg) per kilogram (kg) solution for infusion BI 905677 was administered intravenously on Day 1 of each 3-week treatment cycle. Patients could stay on treatment for unlimited cycles, until disease progression or other criteria for stopping treatment were met.
- BI 905677 0.1 mg/kg: 0.1 milligrams (mg) per kilogram (kg) solution for infusion BI 905677 was administered intravenously on Day 1 of each 3-week treatment cycle. Patients could stay on treatment for unlimited cycles, until disease progression or other criteria for stopping treatment were met.
- BI 905677 0.2 mg/kg: 0.2 milligrams (mg) per kilogram (kg) solution for infusion BI 905677 was administered intravenously on Day 1 of each 3-week treatment cycle. Patients could stay on treatment for unlimited cycles, until disease progression or other criteria for stopping treatment were met.
- BI 905677 0.4 mg/kg: 0.4 milligrams (mg) per kilogram (kg) solution for infusion BI 905677 was administered intravenously on Day 1 of each 3-week treatment cycle. Patients could stay on treatment for unlimited cycles, until disease progression or other criteria for stopping treatment were met.
- BI 905677 0.8 mg/kg: 0.8 milligrams (mg) per kilogram (kg) solution for infusion BI 905677 was administered intravenously on Day 1 of each 3-week treatment cycle. Patients could stay on treatment for unlimited cycles, until disease progression or other criteria for stopping treatment were met.
- BI 905677 1.6 mg/kg: 1.6 milligrams (mg) per kilogram (kg) solution for infusion BI 905677 was administered intravenously on Day 1 of each 3-week treatment cycle. Patients could stay on treatment for unlimited cycles, until disease progression or other criteria for stopping treatment were met.
- BI 905677 2.4 mg/kg: 2.4 milligrams (mg) per kilogram (kg) solution for infusion BI 905677 was administered intravenously on Day 1 of each 3-week treatment cycle. Patients could stay on treatment for unlimited cycles, until disease progression or other criteria for stopping treatment were met.
- BI 905677 2.8 mg/kg: 2.8 milligrams (mg) per kilogram (kg) solution for infusion BI 905677 was administered intravenously on Day 1 of each 3-week treatment cycle. Patients could stay on treatment for unlimited cycles, until disease progression or other criteria for stopping treatment were met.
- BI 905677 3.6 mg/kg: 3.6 milligrams (mg) per kilogram (kg) solution for infusion BI 905677 was administered intravenously on Day 1 of each 3-week treatment cycle. Patients could stay on treatment for unlimited cycles, until disease progression or other criteria for stopping treatment were met.
Period: Overall Study
Arm/Group | BI 905677 0.05 mg/kg | BI 905677 0.1 mg/kg | BI 905677 0.2 mg/kg | BI 905677 0.4 mg/kg | BI 905677 0.8 mg/kg | BI 905677 1.6 mg/kg | BI 905677 2.4 mg/kg | BI 905677 2.8 mg/kg | BI 905677 3.6 mg/kg
Started | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 7 | 3
Completed | 3 | 3 | 3 | 2 | 3 | 5 | 5 | 6 | 1
Not Completed | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Missing visit | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): includes all patients who received at least one infusion of BI 905677.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 905677 0.05 mg/kg | BI 905677 0.1 mg/kg | BI 905677 0.2 mg/kg | BI 905677 0.4 mg/kg | BI 905677 0.8 mg/kg | BI 905677 1.6 mg/kg | BI 905677 2.4 mg/kg | BI 905677 2.8 mg/kg | BI 905677 3.6 mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 7 | 3 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.3 (17.4) | 57.7 (8.0) | 54.7 (10.0) | 58.3 (10.7) | 50.7 (7.6) | 58.3 (11.3) | 55.0 (10.8) | 52.3 (14.9) | 64.0 (2.6) | 55.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 0 | 2 | 4 | 1 | 4 | 1 | 13
  Male | 2 | 3 | 3 | 3 | 1 | 2 | 5 | 3 | 2 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 3 | 3 | 3 | 5 | 6 | 7 | 2 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 1 | 3 | 2 | 2 | 1 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 3 | 2 | 2 | 3 | 2 | 3 | 2 | 5 | 2 | 24
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: The number of participants with Dose Limiting Toxicities (DLTs) is reported. Any of the following adverse events (AEs) will be classified as DLTs following review by the Safety Monitoring Committee and the Medical Monitor, unless unequivocally due to underlying malignancy or an extraneous cause, including any AE which prevents a patient starting Cycle 2 within 14 days of completion of Cycle 1; Bone mineral density change of >5% from baseline, confirmed at least 2 months after initial observation; β-CTX increase of more than two-fold from baseline; Grade 3 osteoporosis, and so on.
Time Frame: In the first treatment cycle, up to 3 weeks
Population: Maximum Tolerated Dose (MTD) Evaluation Set (MTDS): includes all patients in the treated set who were not replaced for the MTD determination.
Measure: Count of Participants; unit: Participants
Arm/Group | BI 905677 0.05 mg/kg | BI 905677 0.1 mg/kg | BI 905677 0.2 mg/kg | BI 905677 0.4 mg/kg | BI 905677 0.8 mg/kg | BI 905677 1.6 mg/kg | BI 905677 2.4 mg/kg | BI 905677 2.8 mg/kg | BI 905677 3.6 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Statistical Analysis 1: Comparison: BI 905677 0.05 mg/kg; Bayesian logistic regression model (BLRM) with overdose control was used to determine the maximum tolerated dose (MTD), defined as highest dose with less than 25% risk of the true DLT rate being equal to or above 33%; Test type: Other; Probability of DLT rate in [0.16, 0.33) = 0 — Posterior probabilities of the DLT rate lying in the intervals [0.16, 0.33) (target dosing), and [0.33,1] (overdosing) are reported; Probability of DLT rate in [0.33, 1] = 0
Statistical Analysis 2: Comparison: BI 905677 0.1 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other; Probability of DLT rate in [0.16, 0.33) = 0 — [estimate comment as in outcome 1, analysis 1]; Probability of DLT rate in [0.33, 1] = 0
Statistical Analysis 3: Comparison: BI 905677 0.2 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other; Probability of DLT rate in [0.16, 0.33) = 0 — [estimate comment as in outcome 1, analysis 1]; Probability of DLT rate in [0.33, 1] = 0
Statistical Analysis 4: Comparison: BI 905677 0.4 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other; Probability of DLT rate in [0.16, 0.33) = 0 — [estimate comment as in outcome 1, analysis 1]; Probability of DLT rate in [0.33, 1] = 0
Statistical Analysis 5: Comparison: BI 905677 0.8 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other; Probability of DLT rate in [0.16, 0.33) = 0 — [estimate comment as in outcome 1, analysis 1]; Probability of DLT rate in [0.33, 1] = 0
Statistical Analysis 6: Comparison: BI 905677 1.6 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other; Probability of DLT rate in [0.16, 0.33) = 0.003 — [estimate comment as in outcome 1, analysis 1]; Probability of DLT rate in [0.33, 1] = 0
Statistical Analysis 7: Comparison: BI 905677 2.4 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other; Probability of DLT rate in [0.16, 0.33) = 0.035 — [estimate comment as in outcome 1, analysis 1]; Probability of DLT rate in [0.33, 1] = 0.001
Statistical Analysis 8: Comparison: BI 905677 2.8 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other; Probability of DLT rate in [0.16, 0.33) = 0.176 — [estimate comment as in outcome 1, analysis 1]; Probability of DLT rate in [0.33, 1] = 0.018
Statistical Analysis 9: Comparison: BI 905677 3.6 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other; Probability of DLT rate in [0.16, 0.33) = 0.129 — [estimate comment as in outcome 1, analysis 1]; Probability of DLT rate in [0.33, 1] = 0.83

2. Primary Outcome: Number of Patients Experiencing Adverse Events (AEs) During the Entire Treatment Period
Description: The Number of patients experiencing adverse events (AEs) during the entire treatment period is reported.
Time Frame: From first dose until last dose + 42 days (6 weeks) of residual effect period, up to 36 weeks.
Population: Treated Set (TS): includes all patients who received at least one infusion of BI 905677.
Measure: Count of Participants; unit: Participants
Arm/Group | BI 905677 0.05 mg/kg | BI 905677 0.1 mg/kg | BI 905677 0.2 mg/kg | BI 905677 0.4 mg/kg | BI 905677 0.8 mg/kg | BI 905677 1.6 mg/kg | BI 905677 2.4 mg/kg | BI 905677 2.8 mg/kg | BI 905677 3.6 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 7 | 3
Participants | 3 | 3 | 2 | 3 | 3 | 6 | 6 | 7 | 3

3. Secondary Outcome: Maximum Measured Concentration of BI 905677 in Serum After First Infusion (Cmax)
Description: The Maximum measured concentration of BI 905677 in serum after first infusion is reported.
Time Frame: 5 minutes (min) before and at 1, 1.5, 4, 8, 24, 72, 168 and 336 hour(s) after first dosing in Cycle 1.
Population: Pharmacokinetics (PK) Analysis Set (PKS): The PK set included all patients in the treated set who provided at least one observation for at least one PK endpoint without important protocol violations relevant to the evaluation of PK. Only participants with non-missing outcomes were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram / milliliter
Arm/Group | BI 905677 0.05 mg/kg | BI 905677 0.1 mg/kg | BI 905677 0.2 mg/kg | BI 905677 0.4 mg/kg | BI 905677 0.8 mg/kg | BI 905677 1.6 mg/kg | BI 905677 2.4 mg/kg | BI 905677 2.8 mg/kg | BI 905677 3.6 mg/kg
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 2 | 6 | 6 | 6 | 3
nanogram / milliliter | 512 (20.7) | 1100 (22.00) | 1720 (6.59) | 4890 (23.1) | 6540 (30.9) | 13700 (25.8) | 23100 (17.6) | 26800 (18.5) | 47500 (17.1)

4. Secondary Outcome: Area Under the Serum Concentration-time Curve Over the Time Interval From 0 to the Last Measured Time Point (AUC0-tz)
Description: The Area under the serum concentration-time curve over the time interval from 0 to the last measured time point is reported.
Time Frame: 5 minutes (min) before and at 1 1.5, 4, 8, 24, 72, 168 and 336 hour(s) after first dosing in Cycle 1.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram * hour / milliliter
Arm/Group | BI 905677 0.05 mg/kg | BI 905677 0.1 mg/kg | BI 905677 0.2 mg/kg | BI 905677 0.4 mg/kg | BI 905677 0.8 mg/kg | BI 905677 1.6 mg/kg | BI 905677 2.4 mg/kg | BI 905677 2.8 mg/kg | BI 905677 3.6 mg/kg
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 2 | 6 | 6 | 6 | 3
nanogram * hour / milliliter | 8260 (64.5) | 26000 (11.00) | 49700 (16.0) | 144000 (66.6) | 258000 (43.7) | 694000 (22.3) | 1130000 (10.6) | 1170000 (30.4) | 1950000 (32.5)

ADVERSE EVENTS:
Time Frame: For adverse events: From first dose until last dose + 42 days (6 weeks) of residual effect period (REP), up to 36 weeks. For all-cause mortality: From first dose through last dose until end of follow-up, up to 30 weeks + 6 months.
Description: Treated Set (TS): includes all patients who received at least one infusion of BI 905677.
Arm/Group | BI 905677 0.05 mg/kg | BI 905677 0.1 mg/kg | BI 905677 0.2 mg/kg | BI 905677 0.4 mg/kg | BI 905677 0.8 mg/kg | BI 905677 1.6 mg/kg | BI 905677 2.4 mg/kg | BI 905677 2.8 mg/kg | BI 905677 3.6 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 0/3 | 1/3 | 1/3 | 0/6 | 2/6 | 1/7 | 1/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 1/3 | 2/3 | 1/3 | 2/6 | 4/6 | 7/7 | 3/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 2/3 | 3/3 | 3/3 | 6/6 | 6/6 | 7/7 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 905677 0.05 mg/kg (N=3) | BI 905677 0.1 mg/kg (N=3) | BI 905677 0.2 mg/kg (N=3) | BI 905677 0.4 mg/kg (N=3) | BI 905677 0.8 mg/kg (N=3) | BI 905677 1.6 mg/kg (N=6) | BI 905677 2.4 mg/kg (N=6) | BI 905677 2.8 mg/kg (N=7) | BI 905677 3.6 mg/kg (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stoma site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood electrolytes decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
C-telopeptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 905677 0.05 mg/kg (N=3) | BI 905677 0.1 mg/kg (N=3) | BI 905677 0.2 mg/kg (N=3) | BI 905677 0.4 mg/kg (N=3) | BI 905677 0.8 mg/kg (N=3) | BI 905677 1.6 mg/kg (N=6) | BI 905677 2.4 mg/kg (N=6) | BI 905677 2.8 mg/kg (N=7) | BI 905677 3.6 mg/kg (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 0 | 4 | 3 | 3 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 3 | 2 | 2 | 2 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 1 | 2 | 3 | 3 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enterocolitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bone density decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
C-telopeptide increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2 | 2 | 3 | 3 | 2 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypotriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Recruitment into Schedule B was planned start after the maximum tolerated dose of Schedule A was reached. Study was terminated prematurely due to sponsor decision before Schedule B starting. The planned Schedule B part was not held.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT03604445/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT03604445/SAP_001.pdf